CLINICAL TRIAL: NCT00955227
Title: Can Cholesterol Lowering Drugs Influence Circulating Omega-3 Fatty Acid Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Grant Pierce, Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: B2009:054
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Hypercholesterolemia; Hyperlipidemia
Keywords: Omega-3 Fatty acid; ALA (alpha linolenic acid); Ezetimibe; Flaxseed oil capsules
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — Linseed Oil; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Statins only (No Intervention): In this arm- 15 Patients with heart disease and hypercholesterolemia will receive standard statin treatment as determined by the Cardiologist. Patients in this arm will be excluded if they are on ezetimibe.
- Statins and ezetimibe (Active Comparator): In this arm- 15 Patients with heart disease and hypercholesterolemia will receive standard statin treatment as determined by the Cardiologist. In addition, these patients will be on ezetimibe.
  Interventions: Drug: Ezetimibe
- Statins and flax oil only (Experimental): In this arm- 15 Patients receiving standard statin treatment as determined by their cardiologist will also receive two flaxseed oil capsules/day each containing 500 mg of ALA.
  Interventions: Dietary Supplement: Flax seed oil (ALA)
- Statins and ezetimibe and flax oil (Experimental): In this arm- 15 Patients with heart disease and hypercholesterolemia that are on standard statin treatment as determined by their cardiologist, will also receive (as an intervention) ezetimibe and flaxseed oil capsules containing 500mg of ALA.
  Interventions: Dietary Supplement: Flax seed oil (ALA); Drug: Ezetimibe

INTERVENTIONS:
Dietary Supplement: Flax seed oil (ALA) — 2 capsules each containing 500mg of ALA will be taken once per day for 6 weeks
  Other Names: Jamieson Flax seed oil (ALA)- capsules.
  Arms: Statins and ezetimibe and flax oil; Statins and flax oil only
Drug: Ezetimibe — In total, 30 patients will receive ezetimibe as a drug intervention. The dosage is 10mg pod for 6 weeks
  Arms: Statins and ezetimibe; Statins and ezetimibe and flax oil

SUMMARY:
The objective of this study is to determine if the administration of a cholesterol lowering drug like ezetimibe will reduce circulating omega-3 fatty acid (ALA) levels in patients with heart disease and hypercholesterolemia.

The investigators hypothesize that their data will discover that patients receiving ezetimibe require additional dietary supplementation with omega-3 supplements to insure that these beneficial fatty acids are available to these patients.

DETAILED DESCRIPTION:
All patients will undergo drug therapy as required to treat their clinical symptoms including the use of other classes of cholesterol-lowering drugs like statins (that will not interfere with intestinal cholesterol levels). One group of patients will be those who in addition to there existing drug therapy are prescribed ezetimibe to lower circulating cholesterol concentrations. A second group of patients will be those who are not prescribed ezetimibe as part of their normal course of therapy. Blood samples will be taken from all patients at the study baseline. All patients will be fasted for 12 hours prior to the blood sample being taken. After 6 weeks a second blood sample will be taken. This will determine if the drug intervention (ezetimibe) influenced the circulating omega-3 fatty acid concentration.

It will also be of interest to determine if drug administration (ezetimibe) will influence this process when higher levels of omega-3 fatty acids are given to the patients by dietary supplements of ALA. Two additional groups of patients will consume a flaxseed oil supplement containing 1g of ALA in the form of two capsules daily

ELIGIBILITY:
Inclusion Criteria:

* The subject is between 18-80 years old
* The subject lives in Winnipeg area
* The subject is willing to seize intake of oils/ salad dressings/ seafood
* The subject is willing to comply with the study schedule

Exclusion Criteria:

* The subject had been taking flax oil in the last month
* The subject is not willing to undergo dietary restrictions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07; Primary Completion 2011-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Levels of circulating omega-3 fatty acid (ALA) | 6 weeks after enrollment of patient

SECONDARY OUTCOMES:
The n6:n3 fatty acid ratio will be calculated Total cholesterol, LDL, HDL, and triglyceride levels will also be measured | 6 weeks after patient enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Grant N Pierce, PhD, Study Director — St. Boniface Hospital; Davinder Jassal, Principal Investigator — St. Boniface Hospital
Locations (2):
- Canada (2):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - St. Boniface General Hospital Research Centre, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: Yes
Results in press in 2016 Clinical Nutrition Blackwood et. al

REFERENCES:
- [Derived] Blackwood DP, LaVallee RK, Al Busaidi A, Jassal DS, Pierce GN. A randomized trial of the effects of ezetimibe on the absorption of omega-3 fatty acids in cardiac disease patients: A pilot study. Clin Nutr ESPEN. 2015 Oct;10(5):e155-e159. doi: 10.1016/j.clnesp.2015.07.002. Epub 2015 Aug 28. PMID 28531469